CLINICAL TRIAL: NCT04665349
Title: Effect of Fasting on the Non-invasive Measurement of the Body's Water Compartments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Clinical Professor, Head of Department of Anaesthesiology and Intensive Care, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NKBBN/126/2014
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Dehydration; Perioperative Complication
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-op (Experimental): Nutricia Pre-op, 400 milliliters, per os
  Interventions: Dietary Supplement: Nutricia Pre-op, 400 milliliters, per os
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Nutricia Pre-op, 400 milliliters, per os — After 10 hours of fasting participants will receive per os 400 milliliters of Nutricia Pre-op
  Arms: Pre-op

SUMMARY:
Preoperative fasting is defined as refraining from food for at least 6 hours and clear fluids for at least 2 hours prior to anaesthesia. On the one hand, it is a procedure that reduces the risk of aspiration of food content and the occurrence of Mendelson's syndrome, and on the other hand, it was considered to be the cause of disturbances in water management in patients undergoing general anaesthesia. However, reports from recent years have found that moderate preoperative fasting does not influence the risk of hypovolemia in anesthetized patients. It is also known that in fasting people the total body water is reduced. Thus, it can be assumed that there are mechanisms causing the movement of extravascular water into the lumen of blood vessels. For several years, the Body Composition Monitor (BCM) device for non-invasive measurement of the volume of individual water compartments of the human body has been available on the market. It allows to determine the volume of total body water, intracellular body water and extracellular body water. It is mainly used during dialysis, but it can also be used in other circumstances that require the determination of the body's hydration status. The principle of this method is based on non-invasive bioimpedance measurement with the use of 4 electrodes placed on two extremities.

The aim of the study is to determine whether there is a fluid shift between the intracellular and extracellular compartments in people undergoing preoperative fasting. Examination of this issue would allow for the development of hypothesis regarding the optimal perioperative fluid therapy. If there was a shift of fluid from the intracellular space, it seems more rational to supplement fluid deficiencies resulting from starvation with a 5% glucose solution. If, on the other hand, no fluid shift from the intracellular space was detected, which would suggest shifts within the extracellular space, it would be advisable to hydrate the patient with crystalloid solutions.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) general condition assessment 1 or 2

Exclusion Criteria:

* Chronic kidney disease
* Circulatory failure
* Phenylketonuria
* History of hypoglycaemic episodes or any carbohydrate metabolism disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Amount of total body water | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Measurements will be done with Fresenius Body Composition Monitor
Extracellular to intracellular water ratio | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Measurements will be done with Fresenius Body Composition Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Owczuk, Professor, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuklinski J, Steckiewicz KP, Sekula B, Aszkielowicz A, Owczuk R. The influence of fasting and carbohydrate-enriched drink administration on body water amount and distribution: a volunteer randomized study. Perioper Med (Lond). 2021 Aug 10;10(1):27. doi: 10.1186/s13741-021-00198-0. PMID 34372928